CLINICAL TRIAL: NCT03413085
Title: A Prospective, Randomization, Double-blind Study to Evaluate the Efficacy and Safety of Multifocal Soft Contact Lens in Myopia Control
Brief Title: To Evaluate the Efficacy and Safety of Multifocal Soft Contact Lens in Myopia Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Largan Medical Co., Ltd. (Industry)
Collaborators: National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LMO00-CL-DM-01
Record Dates: First submitted 2018-01-21; First posted 2018-01-29 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Myopia
Keywords: Myopia control
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Intervention Model Description: Paired-eye comparison
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Intervention name: multifocal soft contact lens/single vision soft contact lens
  Left eye: multifocal soft contact lens Right eye: single vision soft contact lens
  Interventions: Device: soft contact lens
- Group B (Other): Intervention name: multifocal soft contact lens/single vision soft contact lens
  Left eye: single vision soft contact lens Right eye: multifocal soft contact lens
  Interventions: Device: soft contact lens

INTERVENTIONS:
Device: soft contact lens — Group A
  Group B

SUMMARY:
The objective of this study is to investigate the efficacy and safety of soft lens in myopia control.

DETAILED DESCRIPTION:
This is a prospective, randomized, paired eye comparison, double-blind study aims to evaluate the efficacy and safety of "Soft Lens" in myopia control among schoolchildren. A total of 118 eyes are planned to be enrolled and the expect duration of subject participation will be 48 weeks not including two weeks of screening period. Data such as refractive error, axial length, visual acuity, average wearing hours, self-assessment, adverse events etc. will be collected during the study. A total of 10 visits, i.e. a screening visit, a randomization visit, and 8 treatment visits are planned. Subjects will be encouraged to complete all planned visits.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders aged between 6 and 15 years
2. Spherical equivalent refractive error between -1.00D and -10.00D
3. Visual acuity with contact lens of 20/25 or better in each eye
4. Astigmatism less than or equal to 1.50D
5. Anisometropia less than or equal to 1.00D
6. Agree to wear assigned contact lens and able to comply with the study protocol
7. Subjects and/or their legal representatives agree to sign informed consent form

Exclusion Criteria:

1. Eye disease or vision problem that may contraindicate/interfere with contact lens wearing, for example:

   1. Amblyopia
   2. Severe strabismus at investigator's discretion
   3. Pathologically dry eye
   4. Aphakia
   5. Slit lamp findings including but not limited to corneal edema, corneal ulcer, bulbar redness that are more serious than grade 1
   6. Currently ocular infection of any type or inflammation in either eye
   7. Oculomotor nerve palsies
   8. Pupil or lid abnormality in either eye
   9. Severe ocular allergy
   10. Anterior segment infection, inflammation or abnormality
   11. Corneal vascularization greater than 1 mm of penetration
   12. History of herpetic keratitis
2. Use of bifocals, progressive addition lenses, rigid gas permeable contact lenses, orthokeratology lenses, atropine, pirenzepine or any other myopia control treatment within 1 month prior to screening visit
3. Systemic disease that may affect vision or contact lens wearing (e.g. diabetes, Down syndrome), autoimmune disease, infectious disease, or immunosuppressive diseases recorded in medical charts or informed by caregiver
4. Surgically altered eyes (e.g. corneal or refractive surgery, not including stye removal surgery)
5. Receiving any medication for long-term use which may interfere with contact lens wearing, tear film production, pupil size, accommodation or refractive state, such as nasal decongestants (e.g. pseudoephedrine, phenylephrine), antihistamines (e.g. chlorpheniramine, diphenhydramine), Prednisolone or Ritalin (methyphenidate)

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Objective cycloplegic refractive error | 48 weeks
  Changes in objective cycloplegic refractive error between the two eyes in 48 weeks
Axial length | 48 weeks
  Changes in axial length between the two eyes in 48 weeks

SECONDARY OUTCOMES:
Cycloplegic refractive error | 12, 24, and 36 weeks
  Changes in objective cycloplegic refractive error between the two eyes from baseline after treatment
Axial length | 12, 24, and 36 weeks
  Changes in axial length between the two eyes from baseline after treatment
Myopia progression and axial elongation | during 48 weeks
  Percent reductions of myopia progression and axial elongation
Self-assessment by questionnaire 1 | during 48 weeks
  Analysis of subject self-assessment
Self-assessment by questionnaire 2 | during 48 weeks
  Average wearing hours across the study period
Self-assessment by questionnaire 3 | during 48 weeks
  Reasons and rate for discontinued wear during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Hsun Tsai, M.D., Study Chair — National Taiwan University Hospital; Tzu-Hsun Tsai, M.D., Principal Investigator — National Taiwan University Hospital; Chao-Wen Lin, M.D., Principal Investigator — National Taiwan University Hospital; Ken-Kuo Lin, M.D., Principal Investigator — Taipei Chang Gung Memorial Hospital; Jiahn-Shing Lee, M.D., Principal Investigator — Chang Gung Memorial Hospital; Chiun-Ho Hou, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (3):
- Taiwan (3):
  - Tzu-Hsun Tsai M.D., Taipei
  - Ken-Kuo Lin M.D., Taipei
  - Jiahn-Shing Lee M.D., Taoyuan District

IPD SHARING:
Plan to Share IPD: No